CLINICAL TRIAL: NCT05167279
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Clinical Trial to Evaluate the Tolerability, Safety, Pharmacokinetic Profiles, and Immunogenicity of JS026 and JS026 in Together With JS016 Administered Intravenously to Healthy Chinese Subjects
Brief Title: A Study of JS026 and JS026 Together With JS016 for Treatment of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: JS026-001-I
Record Dates: First submitted 2021-12-13; First posted 2021-12-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — JS026; etesevimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- JS026/placebo 30 mg (Placebo Comparator): 4 patients will be enrolled in this arm.
  Interventions: Biological: JS026/placebo; Biological: JS016/placebo
- JS026/placebo 100 mg (Placebo Comparator): 4 patients will be enrolled in this arm.
  Interventions: Biological: JS026/placebo; Biological: JS016/placebo
- JS026/placebo 300 mg (Placebo Comparator): 8 patients will be enrolled in this arm.
  Interventions: Biological: JS026/placebo; Biological: JS016/placebo
- JS026/placebo 600 mg (Placebo Comparator): 8 patients will be enrolled in this arm.
  Interventions: Biological: JS026/placebo; Biological: JS016/placebo
- JS026/placebo 1000 mg (Placebo Comparator): 8 patients will be enrolled in this arm.
  Interventions: Biological: JS026/placebo; Biological: JS016/placebo
- JS026/placebo 300 mg + JS016/placebo1200 mg (Placebo Comparator): 8 patients will be enrolled in this arm.
  Interventions: Biological: JS026/placebo; Biological: JS016/placebo
- JS026/placebo 600 mg + JS016/placebo 1200 mg (Placebo Comparator): 8 patients will be enrolled in this arm.
  Interventions: Biological: JS026/placebo; Biological: JS016/placebo

INTERVENTIONS:
Biological: JS026/placebo — Five dose groups (30 mg, 100 mg, 300 mg, 600 mg, and 1000 mg) will be set to receive an intravenous infusion of JS026/placebo on Day1, and two dose groups (300 mg JS026 + 1200 mg JS016, and 600 mg JS026+ 1200 mg JS016) will be set to receive an intravenous infusion of JS026/placebo + JS016/placebo on Day1. The investigational product and placebo will be distributed in each dose group in a ratio of 3:1.
Biological: JS016/placebo — Two dose groups (300 mg + 1200 mg, and 600 mg + 1200 mg) will be set to receive an intravenous infusion of JS026/placebo + JS016/placebo on Day1. The investigational product and placebo will be distributed in each dose group in a ratio of 3:1.

SUMMARY:
This is a first-in-human (FIH), randomized, double-blind, placebo-controlled, single-center phase I clinical trial of JS026 and JS026 + JS016 Injection. The objective of the study is to evaluate the safety, tolerability, PK profile and immunogenicity of a single intravenous infusion of JS026 and JS026 + JS016 Injection in healthy subjects.

In this study, the single ascending dose design will be adopted, JS026 will be administered sequentially from low dose group to high dose group, and each subject can only receive an intravenous infusion at one dose level. Five dose groups (30 mg, 100 mg, 300 mg, 600 mg, and 1000 mg) will be set to receive an intravenous infusion of JS026, and two dose groups (300 mg JS026 + 1200 mg JS016, and 600 mg JS026+ 1200 mg JS016) will be set for JS026 + JS016. The investigational product and placebo will be distributed in each dose group in a ratio of 3:1. Four subjects will be enrolled in each of JS026 30 mg and 100 mg groups, and 8 subjects will be enrolled in each of other dose groups, totally 48 subjects.

DETAILED DESCRIPTION:
The entire trial period consists of a screening period of up to 14 days, a single dosing day (D1), and a 12-week follow-up period (84 days after dosing). Subjects will be admitted to the phase I clinical trial ward on the day before administration (D-1), and discharged after all examinations and assessments are completed on D4 after administration. Moreover, they will return to thestudy site for follow-up visits and relevant procedures and assessments as scheduled in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects
* Body weight ≥ 50 kg for males and ≥ 45 kg for females
* Female subjects must meet the following criteria: not of childbearing potential (e.g., documented hysterectomy, bilateral salpingectomy or ligation, or more than 1 year of amenorrhea), or of childbearing potential with a negative blood pregnancy test at screening, and willing to take strict and effective contraceptive measures (e.g., abstinence, medication, or barrier method [e.g., contraceptive sponge, vaginal cuff, vaginal diaphragm, cervical cap, etc.]) for 6 months after dosing. Male subjects must agree to take strict and effective contraceptive measures (eg, abstinence, drug, or barrier method [e.g., male condom]) for 6 months after dosing.
* Results of medical evaluations, including physical examination, vital signs, laboratory tests, and other auxiliary examinations (chest imaging, abdominal B ultrasound, ECG, etc.) are normal or abnormal without clinical significance.
* Able to read and understand the contents of the trial, willing to participate in the trial and comply with the trial protocol and procedures, and having signed the written ICF.

Exclusion Criteria:

* Patients with past medical history or current clinically significant concomitant diseases;
* History of malignancies within 5 years.
* Receiving any prescription drugs or over-the-counter drugs, including herbal remedies, vitamins, and dietary supplements, within 14 days prior to screening.
* Participating in any clinical trial with drug intervention within 3 months prior to screening, or the drug is within the elimination phase (5 elimination half-lives), whichever is longer.
* Receiving any therapeutic or investigational biologic within 6 months prior to screening.
* With a history of drug abuse within 1 year, or a positive result at screening.
* Females who are pregnant or lactating.
* Any other condition that the investigator deems inappropriate to participate in the trial, such as subject's mental or legal incapacity, potential compliance problems, and failure to complete the study-related procedures according to the requirements of the protocol, as determined by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence and severity of any adverse events (AEs) occurring during the clinical trial per CTCAE V5.0 | 85 days
  Incidence and severity of any adverse events (AEs) occurring during the clinical trial, including serious adverse events (SAEs), and adverse events of special interest (AESIs), as well as abnormalities in clinical symptoms, vital signs, physical examination, laboratory tests (complete blood cell count, serum chemistry, routine urinalysis, coagulation function, etc.) and 12-lead ECGs will be observed for all the subjects, the their clinical manifestations and features, severity, time to onset, end time, therapeutic measures and outcomes will be recorded, and the correlation of the adverse events with the investigational product will be judged.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | Day 1 to D85
  Area under the plasma concentration-time curve from the time of dosing to the last measurable concentration time t (AUC0-last)
Pharmacokinetics: Tmax | Day 1 to D85
  Time to maximum concentration (Tmax)
Pharmacokinetics: Cmax | Day 1 to D85
  Maximum concentration (Cmax)
Pharmacokinetics: Vd | Day 1 to D85
  Apparent volume of distribution (Vd)
Pharmacokinetics: CLt | Day 1 to D85
  Terminal clearance (CLt)
Pharmacokinetics: t1/2 | Day 1 to D85
  Elimination half-life (t1/2)
Immunogenicity: ADA | Day 1 to D85
  Incidence of anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China